CLINICAL TRIAL: NCT04334317
Title: A Randomized, Double-blind, Placebo-Controlled, 2-Period Crossover, Phase 2 Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral TAK-071 in Parkinson Disease Patients With Cognitive Impairment and an Elevated Risk of Falls
Brief Title: A Study of TAK-071 in People With Parkinson Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-071-2002; U1111-1247-0357 (Other: WHO)
Record Dates: First submitted 2020-03-30; First posted 2020-04-06 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease; Healthy Participants
Keywords: Drug Therapy
MeSH Terms: conditions — Parkinson Disease | interventions — TAK-071

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo + TAK-071 (PD Participants) (Experimental): TAK-071 placebo-matching tablets, orally, once daily for up to first 6 weeks in Period 1, followed by ≥3 weeks washout period, followed by TAK-071 tablets, orally, once daily for up to next 6 weeks in Period 2.
  Interventions: Drug: TAK-071; Drug: Placebo
- TAK-071 + Placebo (PD Participants) (Experimental): TAK-071 tablets, orally, once daily for up to first 6 weeks in Period 1, followed by ≥3 weeks washout period, followed by TAK-071 placebo-matching tablets, orally, once daily for up to next 6 weeks in Period 2.
  Interventions: Drug: TAK-071; Drug: Placebo
- Sentinel Cohort: Placebo (Healthy Participants) (Experimental): A single dose of TAK-071 placebo-matching mg, tablet, orally, on Day 1.
  Interventions: Drug: Placebo
- Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants) (Experimental): A single dose of TAK-071 ≤ 7.5 milligrams (mg), tablet, orally, on Day 1.
  Interventions: Drug: TAK-071

INTERVENTIONS:
Drug: TAK-071 — TAK-071 tablet.
  Arms: Placebo + TAK-071 (PD Participants); Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants); TAK-071 + Placebo (PD Participants)
Drug: Placebo — TAK-071 placebo-matching tablet.
  Arms: Placebo + TAK-071 (PD Participants); Sentinel Cohort: Placebo (Healthy Participants); TAK-071 + Placebo (PD Participants)

SUMMARY:
It is hoped that TAK-071 will help people with Parkinson's disease to walk with better balance. The main aim of the study is to check if there is a difference in how participants walk after treatment with TAK-071. Another aim is to see if it improves how participants think and remember.

At the first visit, the study doctor will check who can take part. Participants who can take part will be picked for 1 of 2 groups by chance.

Both groups will have 2 treatments but in a different order. The treatments are TAK-071 tablets or placebo. In this study, a placebo will look like the TAK-071 but will not have any medicine in it.

One group will take TAK-071 for 6 weeks, have at least a 3-week break, then take a placebo for 6 weeks. The other group will take a placebo for 6 weeks, have at least a 3-week break, then take TAK-071 for 6 weeks. The participants will not know the order of their 2 treatments, nor will their study doctors. This is to help make sure the results are more reliable.

The participants will visit the clinic at the beginning and end of each treatment for a check-up. 14 days after the 2nd treatment, clinic staff will telephone the participants for a final check-up.

DETAILED DESCRIPTION:
The drug being tested in this study is TAK-071. TAK-071 is being tested to treat people with PD who have cognitive impairment and are at risk for falls and who are not concurrently taking acetylcholinesterase inhibitors. The study will look at the efficacy and safety of TAK-071 in participants with PD who take TAK-071 versus placebo.

The study will also evaluate the PK of TAK-071 in healthy participants (sentinel cohort) older than 55 years.

The study will enroll approximately 74 participants. An initial sentinel cohort of 10 healthy participants will be included to estimate age effects. Participants aged 56 to 75 years will be randomly assigned in 3:1 ratio to one of the two treatments:

* Sentinel Cohort: TAK-071 7.5 mg
* Sentinel Cohort: Placebo

Enrolment for participants aged 40 to ≤ 85 years in the main study will start simultaneously with sentinel cohort. Based on PK, safety, and physiologically based PK modelling data from sentinel cohort, dosing will be decided for the remaining participants. Participants with maximum age of 66 to 85 years, inclusive, will be enrolled at a dose of 5 mg, and the dose for subjects aged 40 to 65 years, inclusive, will be 7.5 mg. All participants will be asked to take one tablet at the same time each day throughout the study.

The remaining participants aged 40 years to <=85 years will be randomly assigned in 1:1 ratio to one of two treatment sequences in crossover design:

* TAK-071 + Placebo
* Placebo + TAK-071

The study will be conducted in the United States. The minimum time to participate in this study is approximately 15 weeks. Participants will make multiple visits to the clinic and will have home assessments during the third Week of each 6-week treatment period, and will be contacted by telephone at 14 days after completion of the last period for a follow-up assessment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Is an outpatient of any sex aged between 40 and ≤ 85 years, inclusive, at the time of consent.
2. Has a diagnosis of PD according to Movement Disorders Society (MDS) clinical diagnostic criteria for PD. Participants with DLB (i.e., dementia diagnosed before onset of motor symptoms or up to 1 year after onset of motor symptoms) are also eligible, consistent with MDS clinical diagnostic criteria for PD.
3. Has Hoehn and Yahr stage ≥2 and <4 at the screening visit.
4. Has elevated risk for falls as indicated by at least 1 fall in the last 12 months before the screening visit based on the Fall History Assessment where in the opinion of the investigator the falls were a consequence of PD and are at continued elevated risk of falls per investigator judgment. Investigator judgment on fall risk may be informed by information such as, but not limited to, history, physical examination and/or a score ≥2 on item 3.10 on Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III.
5. Has evidence of cognitive impairment as indicated by a Montreal Cognitive Assessment (MoCA) score between 11 and 26, inclusive and additionally can complete the cognitive assessments at screening (as specified in the study manual).
6. Can walk without aid for 2 minutes while doing serial 3 subtraction (with site staff ensuring participant safety in case of falls). Participants who require aids for walking can be included as long as they can complete the walk test without aid.

Inclusion For Healthy Participants:

1. The participant is a healthy individual of either sex aged between 56 and 75 years, inclusive (for initial set of participant in the sentinel cohort) at the time of consent. Older participants may be enrolled after analysis of data from participants aged 56 to 75 years, inclusive.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Key Exclusion Criteria:

1. Has orthostatic hypotension at screening, as defined as a decline in systolic blood pressure greater than 20 mm Hg or a decrease of 10 mm Hg in diastolic blood pressure on standing measured within 1 minute after being supine for at least 5 minutes.
2. Has dyskinesia of sufficient severity to interfere with digital gait assessments during visits (as defined by Movement Disorders Society - Unified Parkinson's Disease Rating Scale [MDS-UPDRS] section 4.1 "Time spent with dyskinesias" and/or section 4.2 "Functional Impact of Dyskinesias" scores greater than [>] 2), or in the opinion of the investigator the participant's dyskinesia is likely to interfere with the digital gait assessments.
3. Has significant risk factors for seizures (a history of seizures as an adult, a history of brain injury, or other risk factors deemed relevant by the investigator).
4. Is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property, or the participant has attempted suicide within the past year before screening. Participants who have positive answers on item number 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) (based on the past year) before randomization are excluded.
5. Is unwilling or unable to discontinue taking cholinesterase inhibitors and/or moderate or strong cytochrome P-450 3A4 inhibitors or inducers at least 30 days before randomization.

Exclusion For Healthy Participants:

1. Participants has body mass index (BMI) less than 18 or greater than 40.
2. Has significant risk factors for seizures (a history of seizures as an adult, a history of brain injury, or other risk factors deemed relevant by the investigator).
3. The participant is unwilling or unable to discontinue taking cholinesterase inhibitors and/or moderate or strong CYP 3A4 inhibitors or inducers at least 30 days before randomization.
4. The participant is taking warfarin.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (21):
- United States (21):
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - University of California Irvine Medical Center, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - PPD Phase 1 Clinic, Orlando, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - USF Medical Clinic, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Feinberg School of Medicine Northwestern University, Chicago, Illinois
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - Quest Research Institute - Hunt - PPDS, Farmington Hills, Michigan
  - Park Nicollet Health Services, Golden Valley, Minnesota
  - University of Rochester Medicine - Movement Disorders Unit, Rochester, New York
  - Neurology Diagnostics, Inc. - ERG - PPDS, Dayton, Ohio
  - University of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Meridian Clinical Research, Norfolk, Virginia
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Shanbhag NM, Padmanabhan JL, Zhang Z, Harel BT, Jia H, Kangarloo T, Yin W, Dowling AV, Laurenza A, Khudyakov P, Galinsky K, Latzman RD, Simuni T, Weintraub D, Horak FB, Lustig C, Maruff P, Simen AA. An Acetylcholine M1 Receptor-Positive Allosteric Modulator (TAK-071) in Parkinson Disease With Cognitive Impairment: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2025 Feb 1;82(2):152-159. doi: 10.1001/jamaneurol.2024.4519. PMID 39761063
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a39d

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 investigative sites in the United States from 21 October 2020 to 27 February 2023.
Pre-assignment Details: Healthy participants were enrolled in the sentinel cohort of the study to receive TAK-071 and Placebo. Along with the sentinel cohort, participants diagnosed with Parkinson disease were enrolled in one of two sequences to receive treatment with either placebo then TAK-071 in sequence 1, or TAK-071 then placebo in sequence 2.
Groups:
- Placebo Then TAK-071 (PD Participants): TAK-071 placebo-matching tablets, orally, once daily for the first 6 weeks (Period 1), followed by ≥3 weeks washout period, followed by 5 or 7.5 milligrams (mg) TAK-071 tablets - depending on the participant's age orally, once daily for the next 6 weeks (Period 2).
- TAK-071 Then Placebo (PD Participants): Either 5 or 7.5 mg TAK-071 tablets - depending on the participant's age orally, once daily for the first 6 weeks (Period 1), followed by ≥3 weeks washout period, followed by TAK-071 placebo-matching tablets, orally, once daily for the next 6 weeks (Period 2).
- Sentinel Cohort: Placebo (Healthy Participants): A single dose of TAK-071 placebo-matching tablet, orally, on Day 1.
- Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants): A single dose of TAK-071, 7.5 mg tablet, orally, on Day 1.
Period: Overall Study
Arm/Group | Placebo Then TAK-071 (PD Participants) | TAK-071 Then Placebo (PD Participants) | Sentinel Cohort: Placebo (Healthy Participants) | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants)
Started | 26 | 28 | 2 | 8
Completed | 23 | 23 | 2 | 8
Not Completed | 3 | 5 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants who were randomized and receive at least 1 dose of study drug.
Groups:
- Placebo Then TAK-071 (PD Participants): TAK-071 placebo-matching tablets, orally, once daily for the first 6 weeks (Period 1), followed by ≥3 weeks washout period, followed by 5 or 7.5 milligrams (mg) TAK-071 tablets - depending on the participant's age-orally, once daily for the next 6 weeks (Period 2).
- Sentinel Cohort: Placebo (Healthy Participants): A single dose of TAK-071 placebo-matching, tablet, orally, on Day 1.
- Total: Total of all reporting groups
Arm/Group | Placebo Then TAK-071 (PD Participants) | TAK-071 Then Placebo (PD Participants) | Sentinel Cohort: Placebo (Healthy Participants) | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants) | Total
Number analyzed (Participants) | 26 | 28 | 2 | 8 | 64
Age, Continuous [Mean (Full Range); unit: years] | 69.0 [58 to 83] | 70.4 [59 to 81] | 64.5 [61 to 68] | 65.8 [56 to 74] | 67.4 [56 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 5 | 16
  Male | 23 | 22 | 0 | 3 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 2 | 5
  Not Hispanic or Latino | 25 | 26 | 2 | 6 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 1 | 4
  White | 22 | 25 | 1 | 7 | 55
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Weight [Mean (Full Range); unit: kilograms (kg)] | 83.45 [49.4 to 106.0] | 84.63 [66.0 to 121.4] | 72.90 [61.8 to 84.0] | 79.23 [62.1 to 104.8] | 80.05 [49.4 to 121.4]
Height [Mean (Full Range); unit: centimeters (cm)] | 177.42 [157.0 to 190.5] | 174.49 [159.3 to 188.0] | 165.75 [155.5 to 176.0] | 172.63 [164.0 to 180.0] | 172.5 [155.5 to 190.5]
Body Mass Index (BMI) [Mean (Full Range); unit: kilograms per meters square (kg/m^2)] — BMI = weight (kg)/[height (m)]^2
  kilograms per meters square (kg/m^2) | 26.354 [20.04 to 32.11] | 27.813 [22.13 to 39.65] | 26.338 [25.56 to 27.12] | 26.706 [19.71 to 36.00] | 26.80 [19.71 to 39.65]

OUTCOME MEASURES:

1. Primary Outcome: Main Cohort: Change From Baseline in Stride Time (Gait) Variability During a 2-minute Dual-Task Walking Test After 6-week Treatment With TAK-071 Compared With Placebo
Description: Stride time (or gait) is defined as the time elapsed between the first contact of two consecutive footsteps of the same foot and is expressed in seconds. The standard deviation (SD) of the stride time, recorded for each foot during the 2-minutes, is averaged to obtain stride time (gait) variability. The 2-minute walk was performed with and without simultaneous performance of serial 3 subtraction, which adds a cognitive load to the task. Data are reported with and without cognitive load.
Time Frame: Baseline and Week 6 (for each study period)
Population: Pharmacodynamic (PD) analysis set consisted of all participants who received at least 1 dose of study drug and have at least 1 evaluable pharmacodynamic endpoint. Overall number of participants analyzed are the number of participants with data available for analysis. Number analyzed are the number of participants with data available for analysis at given timepoint.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Without Cognitive Load: Placebo; With Cognitive Load: Placebo: TAK-071 placebo-matching tablet, orally, once daily for main cohort.
- Without Cognitive Load: TAK-071: TAK-071, 5 or 7.5 mg tablet, orally, once daily for main cohort.
- With Cognitive Load: TAK-071: TAK-071 5 or 7.5 mg tablet, orally, once daily for main cohort.
Arm/Group | Without Cognitive Load: Placebo | Without Cognitive Load: TAK-071 | With Cognitive Load: Placebo | With Cognitive Load: TAK-071
Number analyzed (Participants) | 47 | 47 | 47 | 45
seconds
  Baseline | 0.0546 (0.03919) | 0.0625 (0.05601) | 0.0930 (0.07743) | 0.0861 (0.06047)
  Week 6: number analyzed (Participants) | 46 | 41 | 46 | 41
  Week 6 | 0.0534 (0.03638) | 0.0607 (0.05666) | 0.0848 (0.07894) | 0.0925 (0.08156)

2. Primary Outcome: Sentinel Cohort, Cmax: Maximum Observed Plasma Concentration for TAK-071 in Healthy Participants
Time Frame: Day 1: pre-dose and Day 2 to 8: post-dose and at multiple time-points (up to approximately 168 hours)
Population: PK analysis set consisted of all participants who received at least 1 dose of TAK-071 and had at least 1 measurable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants)
Number analyzed (Participants) | 8
nanograms per milliliter (ng/mL) | 186 (35.0)

3. Primary Outcome: Sentinel Cohort, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-071 in Healthy Participants
Time Frame: Day 1: pre-dose and Day 2 to 8: post-dose and at multiple time-points (up to approximately 168 hours)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants)
Number analyzed (Participants) | 8
hours | 1.50 [1.00 to 8.00]

4. Primary Outcome: Sentinel Cohort, AUC24: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours for TAK-071 in Healthy Participants
Time Frame: Day 1: Predose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants)
Number analyzed (Participants) | 8
hours*nanograms per milliliter (h*ng/mL) | 3050 (20.7)

5. Primary Outcome: Sentinel Cohort, AUClast: Area Under The Concentration-Time Curve From Time 0 To The Last Quantifiable Concentration in Healthy Participants
Time Frame: Day 1: pre-dose and Day 2 to 8: post-dose and at multiple time-points (up to approximately 168 hours)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants)
Number analyzed (Participants) | 8
h*ng/mL | 11800 (19.2)

6. Primary Outcome: Sentinel Cohort, AUCinf: Area Under The Concentration-Time Curve From Time 0 To Infinity in Healthy Participants
Time Frame: Day 1: pre-dose and Day 2 to 8: post-dose and at multiple time-points (up to approximately 168 hours)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants)
Number analyzed (Participants) | 8
h*ng/mL | 14600 (28.7)

7. Secondary Outcome: Main Cohort: Change From Baseline in Global Cognition Z-score
Description: The global cognition score was calculated as the average of the available z-scores derived from the following individual cognitive tests administered in the cognitive test battery: 'Executive Function' assessed by One Back Test, Modified Groton Maze Learning Test, 'Memory' assessed by One Card Learning Test, International Shopping List Test - Immediate and Delayed Recall Tests, and 'Attention' assessed by Sustained Attention Test and Symbol Digit Modalities Test. Each raw score on the individual tests was converted to a z-score. A global z-score was calculated as an average of the individual z-scores. As the analysis is based on z-scores, there is no minimum or maximum value. An individual z-score of 0 means the observed score is the same as the group mean score at baseline. A positive z-score means the observed score is better (improvement in cognition) than the group mean score at baseline.
Time Frame: Baseline and Week 6 (for each study period)
Population: PD analysis set consisted of all participants who received at least 1 dose of study drug and have at least 1 evaluable pharmacodynamic endpoint. Overall number of participants analyzed are the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Placebo: TAK-071 placebo-matching tablet, orally, once daily for main cohort.
- TAK-071: TAK-071, 5 or 7.5 mg tablet, orally, once daily for main cohort.
Arm/Group | Placebo | TAK-071
Number analyzed (Participants) | 45 | 38
Z-score | -0.059 (0.3671) | 0.208 (0.3940)

8. Secondary Outcome: Main Cohort: Ctrough: Observed Concentration at the End of a Dosing Interval for TAK-071 in Parkinson Disease (PD) Participants
Time Frame: Day 42 of Period 1 and Period 2: pre-dose and at multiple time-points post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- TAK-071: TAK-071, 5 or 7.5 mg, tablet, orally, once daily for main cohort.
Arm/Group | TAK-071
Number analyzed (Participants) | 44
ng/mL | 339 (43.7)

9. Secondary Outcome: Main Cohort, Cmax: Maximum Observed Plasma Concentration for TAK-071 in PD Participants
Time Frame: Day 1 of Period 1 and Period 2: pre-dose and at multiple time-points post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TAK-071
Number analyzed (Participants) | 53
ng/mL | 125 (33.4)

10. Secondary Outcome: Main Cohort: Cmax,ss: Maximum Observed Plasma Concentration at Steady State for TAK-071 in PD Participants
Time Frame: Day 42 of Period 1 and Period 2: pre-dose and at multiple time-points post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TAK-071
Number analyzed (Participants) | 44
ng/mL | 480 (34.4)

11. Secondary Outcome: Main Cohort: AUC24: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours for TAK-071 in PD Participants
Time Frame: Day 1 of Period 1 and Period 2: pre-dose and at multiple time-points post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TAK-071
Number analyzed (Participants) | 53
h*ng/mL | 2360 (32.6)

12. Secondary Outcome: Main Cohort, AUCtau: Area Under the Plasma Concentration-time Curve During a Dosing Interval for TAK-071 in PD Participants
Time Frame: Day 42 of Period 1 and Period 2: pre-dose and at multiple time-points post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TAK-071
Number analyzed (Participants) | 44
h*ng/mL | 9360 (38.3)

13. Secondary Outcome: Main Cohort, Tmax,ss: Time to Reach the Maximum Plasma Concentration (Cmax) at Steady State for TAK-071 in PD Participants
Time Frame: Day 1 of Period 1 and Period 2: pre-dose and at multiple time-points post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-071
Number analyzed (Participants) | 53
hours | 2.10 [1.30 to 12.00]

14. Secondary Outcome: Main Cohort: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-071 in PD Participants
Time Frame: Day 42 of Period 1 and Period 2: pre-dose and at multiple time-points post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-071
Number analyzed (Participants) | 44
hours | 1.75 [1.10 to 6.00]

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form up to 22 days after the last dose of study treatment (up to approximately 148 days)
Description: Safety set consisted of all participants who were randomized and receive at least 1 dose of study drug.
Groups:
- Main Cohort: Placebo (PD Participants): TAK-071 placebo-matching tablet, orally, once daily for main cohort.
- Main Cohort: TAK-071 (PD Participants): TAK-071, 5 or 7.5 mg tablet, orally, once daily for main cohort.
- Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants): A single dose of TAK-071, 5 or 7.5 mg tablet, orally, on Day 1.
Arm/Group | Main Cohort: Placebo (PD Participants) | Main Cohort: TAK-071 (PD Participants) | Sentinel Cohort: Placebo (Healthy Participants) | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/53 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/53 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 2/49 | 5/53 | 2/2 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Cohort: Placebo (PD Participants) (N=49) | Main Cohort: TAK-071 (PD Participants) (N=53) | Sentinel Cohort: Placebo (Healthy Participants) (N=2) | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants) (N=8)
COVID-19 (Infections and infestations) | 1 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Cohort: Placebo (PD Participants) (N=49) | Main Cohort: TAK-071 (PD Participants) (N=53) | Sentinel Cohort: Placebo (Healthy Participants) (N=2) | Sentinel Cohort: TAK-071 7.5 mg (Healthy Participants) (N=8)
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT04334317/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04334317/SAP_001.pdf